CLINICAL TRIAL: NCT02688595
Title: Randomized Controlled Trial on Central Venous Catheterization Techniques in Neonates: Seldinger Versus Modified Seldinger
Brief Title: Central Venous Catheterization Techniques in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1601-108-736
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Catheterization, Central Venous
Keywords: Infant, Newborn; Ultrasonography
MeSH Terms: interventions — Ultrasonography; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seldinger (Experimental): Use a 23 gauge introducer needle for ultrasound-guided central venous catheterization
  Interventions: Device: Ultrasound; Other: General anesthesia
- Modified Seldinger (Experimental): Use a 22 gauge Angiocath Plus catheter for ultrasound-guided central venous catheterization
  Interventions: Device: Ultrasound; Other: General anesthesia

INTERVENTIONS:
Device: Ultrasound — Ultrasound-guided central venous catheterization in internal jugular vein
Other: General anesthesia — Scheduled operation under general anesthesia

SUMMARY:
The purpose of this study is to compare the differences in central venous catheter insertion time, success rate, and complication between the Seldinger and modified Seldinger technique for ultrasound-guided central venous catheterization in neonates.

ELIGIBILITY:
Inclusion Criteria:

* surgery under general anesthesia
* require central venous catheterization

Exclusion Criteria:

* central vein anomaly
* hematoma in central vein
* catheterization site infection

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
First successful central venous catheterization rate | Interval between skin penetration of the needle or angiocatheter and installation of the indwelling catheter, an expected average of 3 minutes

SECONDARY OUTCOMES:
Time to first puncture of central vein | Interval between skin penetration of the needle or angiocatheter and flashback of blood, an expected average of 30 seconds
Time to guide wire insertion | Interval between skin penetration and removal of the needle or angiocatheter after guide wire insertion, an expected average of 90 seconds
Total time to central venous catheterization | Interval between skin penetration of the needle or angiocatheter and installation of the indwelling catheter, an expected average of 3 minutes
Number of central vein puncture trial | up to 5 times, an expected average observation time of 30 seconds
Number of guide wire insertion trial | up to 5 times, an expected average observation time of 90 seconds
First successful central vein puncture rate | Interval between skin penetration of the needle or angiocatheter and flashback of blood, an expected average of 30 seconds
First successful guide wire insertion rate | Interval between skin penetration and removal of the needle or angiocatheter after guide wire insertion, an expected average of 90 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grebenik CR, Boyce A, Sinclair ME, Evans RD, Mason DG, Martin B. NICE guidelines for central venous catheterization in children. Is the evidence base sufficient? Br J Anaesth. 2004 Jun;92(6):827-30. doi: 10.1093/bja/aeh134. Epub 2004 Apr 30. PMID 15121722
- [Background] Song IK, Lee JH, Kang JE, Oh HW, Kim HS, Park HP, Kim JT. Comparison of central venous catheterization techniques in pediatric patients: needle vs angiocath. Paediatr Anaesth. 2015 Nov;25(11):1120-6. doi: 10.1111/pan.12726. Epub 2015 Aug 6. PMID 26248059
- [Derived] Song IK, Kim EH, Lee JH, Jang YE, Kim HS, Kim JT. Seldinger vs modified Seldinger techniques for ultrasound-guided central venous catheterisation in neonates: a randomised controlled trial. Br J Anaesth. 2018 Dec;121(6):1332-1337. doi: 10.1016/j.bja.2018.08.008. Epub 2018 Sep 7. PMID 30442261